CLINICAL TRIAL: NCT03114345
Title: Correlation Between Pressure Differences and Micro-vascularization Changes in Bedridden Paraplegic Patient
Acronym: VASCIP
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Departure of the PhD in charge of the study
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Hill-Rom (Industry); Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 9830
Record Dates: First submitted 2017-03-30; First posted 2017-04-14 (Actual); Last update posted 2021-12-09 (Actual); Status verified 2021-12

CONDITIONS: Pressure Ulcer; Bedsore; Spinal Cord Injury; Paraplegia
Keywords: Pressure ulcer; Interface pressure; Pressure mapping device; Monitoring; Microvascularization
MeSH Terms: conditions — Pressure Ulcer; Spinal Cord Injuries; Paraplegia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm (Other): Measurement of interface pressure and Measurement of micro-vascularization related parameters
  Interventions: Other: Measurement of interface pressure; Other: Measurement of micro-vascularization related parameters

INTERVENTIONS:
Other: Measurement of interface pressure — A capacitive pressure mapping device (XSensor) is set up on the patient air mattress bed. It records the interface pressure on the whole patient body with one frame every second during one hour. Then the file is saved and the pressure mapping device is removed from the patient hospital bedroom.
Other: Measurement of micro-vascularization related parameters — A medical device called O2C, measuring micro-vascularization related parameters (oxygen saturation, hemoglobin quantity and blood flow) is used. The probe (= an optic fibre) is set up lightly on the patient skin or on a transparent adhesive for 1 minute. The median value of the local micro-vascularization parameters are saved on the O2C interface. The location of the measurement is chosen using the pressure mapping device to locate peak pressure area. Then the O2C is removed from the patient hospital bedroom.

SUMMARY:
Paraplegic patients have defective wound healing for sore below the level of spinal lesion. Defect of vascularization of the healing zone certainly participate to this effect. Therefore, this study want to measure, in a clinical settings, the interface pressure (e.g. the pressure between the patient body and the surface he/she is lying on) to assess the correlation between mechanical stress in term of pressure applied over time and tissue oxygenation which represent micro-vascular function. The aim of this clinical trial is to correlate the variations of pressure intensities and changes in micro-vascularization. The measure are recorded when paraplegic patient came into the hospital for pressure ulcer related surgery. The patient is laying on his/her mattress on top of a flexible pressure mapping device. The micro-vascularization parameters are measured at the area displaying the peak pressure a few minutes after the beginning of the pressure interface recording and one hour later at the same area. The data generated during this monocentric study will help to achieve a better understanding of the relation between pressure and micro-vascularization. In the mid term, it will provide a better and more patient adapted pressure ulcer prevention.

ELIGIBILITY:
Inclusion Criteria:

* Educated consent signed,
* Older than 18,
* Paraplegia for at least 6 months,
* Surgery planned for pressure ulcer resection,

Exclusion Criteria:

* Dementia,
* Stade IV arteritis non-revascularisable,
* Patient with no health insurance,
* Pregnant women or breast-feeding, patient unable to give his or her educated consent, ward of the state (art. L.1121-6, L.1121-7, L.1211-8, L.1211-9),
* Patient taking part in another study which could impact the local micro-vascularization.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2017-11-22 (Actual); Primary Completion 2019-11-22 (Actual); Study Completion 2019-11-22 (Actual)

PRIMARY OUTCOMES:
Measure of the pressure intensity in one area | Measurements are done the same date as the inclusion, during the patient hospitalization for his/her pressure ulcer related surgery.
  Pressure intensity is recorded using a mapping pressure device (XSensor), set up on the patient hospital bed. Hemoglobin quantity is measured the same day, at a precise area identified on the pressure mapping device (peak pressure), using the O2C - a micro-vascularization device. All measure are non-invasive.
Measure of the hemoglobin quantity in the same area | Measurements are done the same date as the inclusion, during the patient hospitalization for his/her pressure ulcer related surgery.
  Hemoglobin quantity is measured the same day, at a precise area identified on the pressure mapping device (peak pressure), using the O2C - a micro-vascularization device. All measure are non-invasive.

SECONDARY OUTCOMES:
Measure of other micro-vascularization related parameters (such as the oxygen saturation and the blood flow) recorded at the same area. | Measurements are done the same date as the inclusion, during the patient hospitalization for his/her pressure ulcer related surgery.
  All micro-vascularization related parameters are measured the same day, at a precise area identified on the pressure mapping device (peak pressure), using the O2C - a micro-vascularization device. All measure are non-invasive.

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Matecki, M.D., Principal Investigator — CHU de Montpellier
Locations (1):
- University Regional Hospital Lapeyronie, Montpellier, Languedoc-Roussillon, France

IPD SHARING:
Plan to Share IPD: No